CLINICAL TRIAL: NCT06765629
Title: Safety and Efficacy of Transcutaneous Tibial Nerve Stimulation in Children With Overactive Bladder: A Prospective, Multicenter, Single-Arm Study
Brief Title: Transcutaneous Tibial Nerve Stimulation Therapy in Children With Overactive Bladder
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University (Unknown)
Responsible Party: Principal Investigator, Qibo Hu, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-IRB-0074-P-01
Record Dates: First submitted 2024-12-31; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-invasive Percutaneous Tibial Nerve Stimulation (TTNS) group (Experimental)
  Interventions: Device: Non-invasive Percutaneous Tibial Nerve Stimulation (TTNS) group

INTERVENTIONS:
Device: Non-invasive Percutaneous Tibial Nerve Stimulation (TTNS) group — After obtaining informed consent from the subjects, the researchers screen the subjects based on the inclusion and exclusion criteria. The wearable non-invasive percutaneous tibial nerve stimulator is placed on the area where the tibial nerve runs at the medial malleolus of the subjects. Once the wearable stimulator is properly fitted, stimulation parameter programming and treatment record management are conducted through the programming software running on the mobile phone.

SUMMARY:
Overactive bladder (OAB) is a syndrome characterized by urinary urgency, often accompanied by frequency and nocturia, with or without urge incontinence, without urinary tract infection or other clear pathological changes. The prevalence of OAB ranges from 9% to 43% in women and 7% to 27% in men, severely affecting patients' quality of life and mental health. Traditional treatments for OAB include behavioral therapy (bladder retraining, pelvic floor muscle training, etc.) and drug therapy (including anticholinergic, antispasmodic drugs, and tricyclic antidepressants, etc.); for refractory overactive bladder syndrome, surgical interventions include bladder augmentation and urinary diversion, etc. However, due to serious complications, lack of efficacy, or significant trauma, these methods are greatly limited in clinical application.

In recent years, with the continuous development of neuromodulation technology, neurostimulation has gradually been applied in the treatment of lower urinary tract dysfunction. Compared with traditional treatments, it does not have side effects such as dry mouth, constipation, blurred vision, etc., and compared with surgical treatment, it reduces side effects such as bleeding and infection. Among them, Tibial Nerve Stimulation (TNS) has become an optional therapy for OAB treatment due to its non-surgical nature, convenience, low risk, high safety, significant efficacy, and relative cost-effectiveness.

With the continuous development of technology, and in order to reduce the invasiveness of treatment, improve safety and convenience, Percutaneous Tibial Nerve Stimulation (PTNS) is gradually shifting towards non-invasive Percutaneous Tibial Nerve Stimulation (TTNS). The main difference between the two is that the former uses fine needle electrodes, while the latter mostly uses surface electrodes, which deliver electrical power to the tibial nerve through skin and soft tissue. Studies have shown that TTNS has the same efficacy as drug therapy, is more effective for OAB symptoms than behavioral interventions, and there is no statistically significant difference in efficacy between TTNS and PTNS. It is recommended as an option to improve OAB by the "European Association of Urology Guidelines on Female Non-neurogenic LUTS (2023)" and the "Chinese Guidelines on Diagnosis and Treatment of Urology and Male Diseases (2022)".

However, there is still a lack of large-scale prospective studies on the use of TTNS for OAB in Asian populations, and most existing studies have observation periods of 3 months or less, lacking high-quality research evidence for long-term efficacy. Therefore, a prospective, multicenter, single-arm study is planned to verify the long-term efficacy of percutaneous tibial nerve stimulation in the treatment of OAB in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with OAB according to the "Chinese Urology and Male Disease Diagnosis and Treatment Guidelines" 2022 edition;
2. Age between 6 and 18 years, gender unrestricted;
3. Need to receive and consent to TTNS treatment for medical reasons;
4. Urination diary (3 days prior to random enrollment) shows an average of ≥8 urination times per 24 hours;
5. The patient or their representative understands the purpose and requirements of this study and signs the informed consent form (if the subject is <8 years old, written consent from the legal guardian is required; if the subject is 8 years old ≤ subject ≤ 18 years old, written informed consent from both the subject and the legal guardian is required); If not co-administering β3 agonists/non-selective β-agonists or anticholinergic drugs during the study period, the medication must be discontinued for at least 7 days before the screening period. If continuing to take β3 agonists/non-selective β-agonists or anticholinergic drugs during the study period, the dosage and method of administration must remain unchanged until the study is completed.

Exclusion Criteria:

1. Those with an implanted pacemaker or implantable cardioverter-defibrillator;
2. Patients with concomitant urinary system diseases: deformities, tumors, obstructions, stones, urinary retention;
3. Patients with stress urinary incontinence and other related diseases affecting urine generation and excretion;
4. Individuals with cognitive impairment, Parkinson's disease, or complete spinal cord injury;
5. Patients with psychiatric disorders who cannot cooperate with medical staff;
6. Patients with pelvic organ prolapse at stage III or higher;
7. Patients who do not have sufficient compliance to cooperate with the treatment and are unable to complete the questionnaires and data collection during the treatment period;
8. Pregnant women or those planning to become pregnant during the study period;
9. Patients who are participating in other clinical studies;
10. Other situations deemed unsuitable for inclusion by the researcher.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-09 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
72-hour Voiding Diary | A month after treatment；Two months after treatment；Three months after treatment；Half year after treatment；One year after treatment

SECONDARY OUTCOMES:
Overactive bladder syndrome score (OABSS) | A month after treatment；Two months after treatment；Three months after treatment；Half year after treatment；One year after treatment
  The minimum value is 0 and the maximum value is 15. 3≤score≤5: Mild OAB 6≤score≤11: Moderate OAB score≥12: Severe OAB
Patient Perception of Bladder Condition Score (PPBC-S) | A month after treatment；Two months after treatment；Three months after treatment；Half year after treatment；One year after treatment
  The score ranges from 1 to 6, with a higher score indicating a more severe impact of bladder symptoms on quality of life.
American Urological Association-Symptom Index-Quality of life (AUA-SI-QOL) | A month after treatment；Two months after treatment；Three months after treatment；Half year after treatment；One year after treatment
  The score is from 0 to 6, with higher scores indicating worse quality of life.
Self-Rating Anxiety Scale (SAS) | A month after treatment；Two months after treatment；Three months after treatment；Half year after treatment；One year after treatment
  The Anxiety Self-Rating Scale involves subjectively evaluating 20 questions. Each question is rated on a frequency scale from 1 to 4, where:
  1. point indicates none or very rarely;
  2. points indicate sometimes;
  3. points indicate most of the time;
  4. points indicate almost always or always.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China